CLINICAL TRIAL: NCT07175610
Title: The LUNET Project: the Italian Systemic Erythematous Lupus Network and Registry
Brief Title: LUpus Eritematoso Sistemico NETwork and Registry
Acronym: LUNET
Status: Not yet recruiting | Type: Observational
Sponsor: Società Italiana di Allergologia, Asma e Immunologia Clinica (Other)
Responsible Party: Sponsor
Other Study IDs: 5
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematous (SLE)
Keywords: Systemic Erythematosus Lupus; Connective Tissue Diseases; Autoimmune Diseases; mmune System Diseases; Biologic Therapies
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The LUNET Registry is intended to serve as a comprehensive primary data source, capturing real-world longitudinal clinical information, and the heterogeneity of patient presentations that are often underrepresented in traditional clinical trials. Ultimately, the LUNET Registry will help to optimize SLE management in routine clinical practice by enabling the compilation of real-world evidence to inform clinical decision-making and health policy. Patients will be enrolled by secondary and tertiary care centres for SLE across Italy in a real-world clinical set-up.

DETAILED DESCRIPTION:
The LUNET's specific objectives are as follows:

* Planning and conducting epidemiological studies to evaluate the incidence and prevalence rates of different clinical manifestations of SLE, and to evaluate short- and long-term outcomes, including survival rates and organ dysfunction, injury, and failure
* Promoting multicenter studies that will compare different patient subgroups based on clinical phenotypes and organ involvement, to attain insights regarding disease expression and progression
* Describing the profile of patients with lupus nephritis in the national population, to improve guidelines on its systematic and standardized assessment.
* Evaluating the presence of central and peripheral nervous system involvement in the national population of patients with SLE, assessing the type, frequency, and severity of neurological symptoms and objective signs, as well as the instrumental techniques used in clinical practice (e.g., Magnetic Resonance Imaging (MRI)
* Assessing biomarker data to support early diagnosis and guide treatment choices
* Improving screening techniques for early identification of organ damage in SLE patients
* Improving early treatment strategies
* Tracking adherence and response to therapy
* Evaluating the short- and long-term real-life effectiveness and safety of old and novel drugs approved for SLE, overall and in groups of patients with specific phenotypes
* Assessing SLE patients' quality of life according to clinical phenotype and treatment approach
* Assessing how socioeconomic status impacts patients' access to healthcare and absenteeism in relation to the disease and various therapeutic approaches
* Evaluating how different therapeutic strategies impact hospitalization
* Assessing the influence of old and novel therapies on fertility, pregnancy, and breastfeeding
* Monitoring cardiovascular risk in SLE patients by evaluating the associated comorbidities, prospective development of cardiovascular events, and biomarker levels (e.g., fasting blood glucose, hemoglobin A1c, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides and pro-BNP)
* Evaluating bone metabolism in patients with SLE through assessment of laboratory measurements (e.g., vitamin D, calcium, phosphorus, calcinuria, and phosphaturia) and instrumental assessments, such as dual-energy X-ray absorptiometry (DEXA) scans
* Monitoring the causes of death among SLE patients

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* confirmed SLE diagnosis according to the SLICC 2012 and/or ACR/EULAR 2019 classification criteria;
* provision of signed written informed consent prior to participation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with SLE according to the SLICC 2012 and/or ACR/EULAR 2019 classification criteria
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission | Every year to ten year
  Number of patients who achieved complete clinical remission or low disease activity
Disease activity | Every year to ten year
  Changes in disease activity (SLEDAI-2k)

CONTACTS AND LOCATIONS:
Overall Officials: Amato de Paulis, Study Chair — Division of Internal Medicine and Clinical Immunology, Center for Basic and Clinical Immunology Research (CISI), University of Naples Federico II, Naples, Italy
Locations (16):
- Italy (16):
  - SOD Clinica Medica, Dip. Medicina Interna- Ospedali Riuniti Marche-AOU delle Marche, Ancona
  - Medicina Interna Universitaria (Guido Baccelli) Azienda Ospedaliera Policlinico Consorziale, Bari
  - U.O. di Medicina, Ospedale Civile "Santa Maria della Sapienza", Battipaglia
  - Allergologia e Immunologia Clinica, Azienda Ospedaliero-Universitaria di Cagliari, Cagliari
  - Struttura organizzativa Dipartimentale Complessa Immunologia e Terapie Cellulari, A.O.U. Careggi, Florence
  - Struttura complessa Allergologia Immunologia Clinica e Reumatologia.Azienda Socio Sanitaria Territoriale di Mantova, Mantova
  - Unità di Immunologia, Reumatologia, Allergologia e Malattie Rare all'IRCCS Ospedale San Raffaele di Milano, Milan
  - Division of Internal Medicine and Clinical Immunology, Azienda Ospedaliera Universitaria Federico II, Napoli
  - SYNERGO - Institute of Clinical Immunotherapy and Advanced Biological Treatmets-Casa di Cura Pierangeli S.r.l., Pescara
  - UO Immunoallergologia clinica, Azienda Ospedaliero Universitaria Pisana, Pisa
  - UOC di Medicina Interna e Nutrizione Clinica -Policlinico Umberto I, Roma
  - Reumatologia e Immunologia Clinica, Humanitas Research Hospital, Rozzano
  - UOC Clinica Immunologica e Reumatologica, A.O.U. San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - SC (U.C.O.) Medicina Clinica Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI), Trieste
  - SCDU Immunologia e Allergologia AO Ordine Mauriziano, University of Turin, Turin
  - Medicina Interna B - Azienda Ospedaliera Universitaria Integrata, Verona

REFERENCES:
- [Background] Mormile I, Brussino L, Canonica GW, Cortini F, Costantino MT, Dagna L, Del Giacco S, Della Casa F, Di Gioacchino M, Emmi G, Moroncini G, Negrini S, Pacella D, Parronchi P, Patella V, Rossi FW, Sirena C, Triggiani M, Vacca A, de Paulis A. The LUNET Project: Developing the Italian Systemic Erythematous Lupus Network. J Clin Med. 2025 Sep 2;14(17):6197. doi: 10.3390/jcm14176197. PMID 40943959